CLINICAL TRIAL: NCT01973309
Title: A Phase 1b Dose Escalation Study of Vantictumab (OMP-18R5) in Combination With Paclitaxel in Patients With Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Vantictumab (OMP-18R5) in Combination With Paclitaxel in Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18R5-002
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Locally Recurrent; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vantictumab combined with paclitaxel (Experimental): Drug: vantictumab combined with paclitaxel - administered intravenously
  Interventions: Drug: Vantictumab combined with paclitaxel

INTERVENTIONS:
Drug: Vantictumab combined with paclitaxel — Vantictumab combined with paclitaxel will be administered IV.
  Other Names: (OMP-18R5)

SUMMARY:
This is an open-label Phase 1b dose-escalation study to assess the safety, tolerability, and PK of vantictumab when combined with paclitaxel.

DETAILED DESCRIPTION:
Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined, up to 10 patients may be enrolled in the cohort-expansion phase to better characterize the safety, tolerability and PK of vantictumab combined with paclitaxel. Up to approximately 34 patients may be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Histologically documented adenocarcinoma of the breast with locally recurrent or metastatic disease

  o Patients with breast cancer overexpressing HER2 are not eligible.
* Availability of tumor tissue, either archival FFPE or obtained at study entry through fresh biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* All acute treatment-related toxicity from prior therapy must have resolved to Grade ≤ 1 prior to study entry
* Adequate hematologic and end-organ function
* Evaluable or measurable disease per RECIST v1.1
* For women of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

* Known significant dose delays during prior treatment with a taxane due to drug-related toxicities
* Prior treatment with more than two regimens of systemic cytotoxic chemotherapy for locally recurrent or metastatic disease
* Treatment with any anti-cancer therapy within 3 weeks prior to initiation of study treatment

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of vantictumab in combination with paclitaxel in patients with locally recurrent or metastatic breast cancer | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-28 days).
  The maximum tolerated dose (MTD) will be determined in patients treated with vantictumab in combination with paclitaxel

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of vantictumab when administered in combination with paclitaxel to patients with locally recurrent or metastatic breast cancer | Plasma sample for Pharmacokinetics (PK) analysis to be obtained prior to the vantictumab infusion on Days 0, 14, 56 and 70 and at the end of the vantictumab infusion with paclitaxel infusion on Days 0 and 56.
  Apparent half life, AUC, clearance, volume of distribution

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center/ Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Tyler, Tyler, Texas

REFERENCES:
- [Derived] Diamond JR, Becerra C, Richards D, Mita A, Osborne C, O'Shaughnessy J, Zhang C, Henner R, Kapoun AM, Xu L, Stagg B, Uttamsingh S, Brachmann RK, Farooki A, Mita M. Phase Ib clinical trial of the anti-frizzled antibody vantictumab (OMP-18R5) plus paclitaxel in patients with locally advanced or metastatic HER2-negative breast cancer. Breast Cancer Res Treat. 2020 Nov;184(1):53-62. doi: 10.1007/s10549-020-05817-w. Epub 2020 Aug 14. PMID 32803633